CLINICAL TRIAL: NCT05695326
Title: Effects of a 3D Printing Technology Learning Program for Rehabilitation Professionals: a Randomized Control Trial
Brief Title: Effects of a 3D Printing Technology Learning Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gunma PAZ College (Other)
Responsible Party: Principal Investigator, Ken Kondo, Assistant professor, Gunma PAZ College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PAZ22-2-1
Record Dates: First submitted 2023-01-05; First posted 2023-01-25 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Educational Problems

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effects of a 3D Printing Technology Learning Program (Experimental)
  Interventions: Behavioral: 3D printing technology learning program

INTERVENTIONS:
Behavioral: 3D printing technology learning program — The study is aimed to evaluate a 3D printing technology learning program for rehabilitation professionals

SUMMARY:
3D printing technology helps rehabilitation professionals make an order-made assistive device (AD). However, most have not learned how to use the technology for clinical practice. The study is aimed to evaluate a 3D printing technology learning program for rehabilitation professionals. Eligible participants who have a licence for physical, occupational or speech-language therapy and have not experienced learning any 3D printing technology. The learning program was conducted in accordance with Kolb's Experiential Learning Theory (Morris TH, 2020). The program was conducted over eight weeks. The outcome measure included the Japanese version of the modified Technology Acceptance Model questionnaire (TAM-J). It consists of 13 items and four scales; Perception of usefulness (28 points total), Perception of ease of use (35 points total), Attitude toward use (14 points total) and Intention to use (14 points total). Within-group analyses were performed using the Wilcoxon signed-rank test for the TAM-J between different time points.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants who have a licence for physical, occupational or speech-language therapy

Exclusion Criteria:

* Participants who have experienced learning any 3D printing technology.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
The Japanese version of modified Technology Acceptance Model questionnaire | Change from Baseline a score of the Japanese version of modified Technology Acceptance Model questionnaire at 2 months
  A higher score means the strong acceptance of 3D printing technology(score range is 13 to 91 points)

CONTACTS AND LOCATIONS:
Locations (1):
- shonan keiiku Hospital, Fujisawa, Kanayama, Japan

IPD SHARING:
Plan to Share IPD: No